CLINICAL TRIAL: NCT04889053
Title: Prospective Cohort Study of Coronary Artery Calcification in Type 2 Diabetes Mellitus (USCAC Study)
Brief Title: Coronary Artery Calcification in Type 2 Diabetes Mellitus (USCAC Study)
Status: Recruiting | Type: Observational
Sponsor: University of South China (Other)
Responsible Party: Sponsor
Other Study IDs: USC-4310T2DMCAC
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes; Vascular Calcification; Coronary Artery Calcification; Strains; Epidemiology; microRNA
Keywords: Type 2 Diabetes; Vascular calcification; Epidemiology; microRNA-32
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vascular Calcification; Sprains and Strains

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- D2M, Vascular calcification-free: Meet the inclusion criteria, there is no calcification detected by low dose prospectively triggered sequential dual-source CT coronary angiography
- D2M with vascular calcification: Meet the inclusion criteria, and have coronary artery calcification ( be confirmed by low dose prospectively triggered sequential dual-source CT coronary angiography)

SUMMARY:
Coronary artery calcification (CAC) is a common complication of type 2 diabetes mellitus(T2DM), which can significantly increase all-cause mortality and the incidence of serious cardiovascular events, and increase the burden of the national economy. The epidemiological characteristics and the clinical progress of CAC are still not clear. Moreover, the pathogenesis of CAC has not yet been fully elucidated, and lack of specific diagnostic indicators. Arterial calcification is an active, reversible, and multifactorial biological process like bone formation. It is generally believed that early detection of calcification lesions and active targeted treatment may be the key to prevention and treatment of vascular calcification. In addition, statins are commonly used in patients with dyslipidemia and can stabilize CAC plaque. However, the timing, dosage and effect of statins are controversial. Moreover, our previous study found that the expression of miR-32 is significantly elevated in patients with CAC, and can promoting vascular calcification. Herein, this study is to conduct a prospective cohort study on T2DM patients with CAC in Hunan province through a multidisciplinary and multi-center cooperation model, the main research objectives include the following three parts: ① To identify the prevalence, incidence, and characteristics of CAC in T2DM patients in Hunan province, and to build a risk assessment model. ② To observe the effects of statins on the occurrence and development of CAC in patients with T2DM, and to provide clinical data for the improvement of medication guidelines; ③To observe the dynamic changes of serum miR-32 in the progression of CAC in patients with T2DM, and to explore its possibility as a serological diagnosis or prognostic bio-maker of CAC. The completion of this research project is expected to bring a new breakthrough in the field of early diagnosis, prognosis evaluation, and intervention treatment of patients with T2DM combined with CAC, and provide an important reference for the formulation of cardiovascular disease prevention and control strategy.

DETAILED DESCRIPTION:
The prospective cohort study of type 2 diabetes mellitus(T2DM) with coronary artery calcification (CAC) is a multi-center, observational clinical study. The study included a baseline survey and 8-year follow-up survey of hospitalized patients with T2DM in seven third-class hospital in Hunan Province (the follow-up is divided into two stages, the first stage is the first 4 years, and the second stage is the last 4 years). The first phase is conducted in three affiliated hospitals of University of South China in Hengyang City, Hunan Province, and the second phase is conducted in four representative Grade-A hospitals according to the geographical location of Hunan Province. The sample size of each center is set to be at least 200 cases, and that of a single center is at most 500 cases. The diagnosis of T2DM is made according to the criteria of the WHO in 1999, and the hyperglycemia caused by type 1 diabetes, gestational diabetes, special type diabetes and other factors are excluded. The volume and density of coronary artery calcification are evaluated by low dose prospectively triggered sequential dual-source CT coronary angiography. The coronary artery calcification score (CACS) is calculated by CAS coring software. MiR-32 is detected by PCR. All in all, this clinical trial is aiming to establishing a prospective long-term follow-up cohort of patients with T2DM complicated with CAC in Hunan Province, to observing the effect of statins on the occurrence and development of CAC in patients with T2DM, and to exploring the dynamic changes of serum miR-32 in this process to determine whether it can be used as an early diagnosis and prognostic marker of vascular calcification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Type 2 diabetes is diagnosed according to WHO diagnostic criteria
* Low dose prospectively triggered sequential dual-source CT coronary angiography can be performed at baseline investigation
* Those subjects are able to understand the purpose and procedure of this study and sign the informed consent voluntarily

Exclusion Criteria:

* Those have received coronary artery stenting or coronary artery bypass grafting
* Those with severe lung (respiratory failure), liver (ALT or AST 3 times normal value or bilirubin increase), renal dysfunction[GFR < 45ml/(min.1.73m2) or dialysis patients
* Malignant tumor
* Mental illness or mental retardation
* Pregnant or lactating women or those with fertility planning
* Concomitant diseases (hyperparathyroidism, sarcoidosis, amyloidosis) affecting calcium balance and soft tissue calcification
* Contraindications of contrast agents
* Based on the judgment of the researcher, the compliance is poor and the study could not be completed according to the requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective cohort study of type 2 diabetes mellitus with coronary artery calcification is a multicenter, observational clinical study for patients with type 2 diabetes mellitus. The study included a baseline survey and an 8-year follow-up survey of hospitalized patients with type 2 diabetes mellitus in seven third-class hospital in Hunan Province. The first phase is conducted in three affiliated hospitals of University of South China in Hengyang City, Hunan Province, and the second phase is conducted in four representative Grade-A hospitals according to the geographical location of Hunan Province. The sample size of each center is set to be at least 200 cases, and that of a single-center is at most 500 cases.
Sampling Method: Non-Probability Sample
Enrollment: 1400 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence and incidence rate of CAC in T2DM | Anticipate completed in December 2026
  Based on the baseline data of cohort study, the prevalence of CAC in hospitalized patients with T2DM in Hunan Province is determined by descriptive analysis, and the characteristics of different gender, age group, degree of obesity and duration of diabetes mellitus are explored. Based on prospective cohort data, the incidence rate and characteristics of CAC in T2DM inpatients in Hunan province of China are defined.

SECONDARY OUTCOMES:
The dynamic changes of miR-32 in the occurrence and development of CAC in patients with T2DM, and to clarify the value of miR-32 as a risk marker for early diagnosis and prognosis of CAC | Anticipate completed in December 2030
  Based on the blood sample of patients in this cohort study, the serum miR-32, OPG and alkaline phosphatase(ALP) are detected by RT-PCR, ELISA and colorimetry at baseline. The low dose prospectively triggered sequential dual-source CT coronary angiography image results are taken as the gold standard, The diagnostic value, sensitivity and specificity of the three indicators in the occurrence of CAC in type 2 diabetes mellitus are analyzed.
The effect of statins on the occurrence and development of CAC in patients with T2DM | Anticipate completed in December 2030
  Based on the observational data of prospective cohort study, the effects of different types, doses and application timing of statins on the progression of CAC and cardiovascular events are studied by analysis of covariance or chi square test

CONTACTS AND LOCATIONS:
Overall Officials: Liu Jianghua, PhD, Study Chair — The First Affiliated Hospital of University of South China
Locations (1):
- The First Affiliated Hospital of University of South China, Hengyang, China

IPD SHARING:
Plan to Share IPD: No